CLINICAL TRIAL: NCT05677789
Title: Defining COVID-19 Infection Severity on Presentation to Hospital: a Multicentre Prospective Study
Brief Title: Defining COVID-19 Infection Severity on Presentation to Hospital
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CORMB-65
Record Dates: First submitted 2023-01-04; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: COVID-19; Infections; Morality; Death, Assisted
MeSH Terms: conditions — COVID-19; Infections; Suicide, Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Participants The patient's CORMB score is 0 to 2: Participants The patient's CORMB score is 0 to 2
  Interventions: Diagnostic Test: Medical observation
- Participants The patient's CORMB score is 3 to 4: Participants The patient's CORMB score is 3 to 4
  Interventions: Diagnostic Test: Supportive treatment (BSC)
- Participants The patient's CORMB score is 5 or above: Participants The patient's CORMB score is 5 or above
  Interventions: Diagnostic Test: Intensive care management

INTERVENTIONS:
Diagnostic Test: Medical observation — Likely suitable for home treatment
  Groups: Participants The patient's CORMB score is 0 to 2
Diagnostic Test: Supportive treatment (BSC) — Consider hospital supervised treatment
  Groups: Participants The patient's CORMB score is 3 to 4
Diagnostic Test: Intensive care management — Manage in hospital as severe pneumonia
  Groups: Participants The patient's CORMB score is 5 or above

SUMMARY:
In the assessment of severity in coronavirus disease 2019 (COVID-19), the modified Brit_x0002_ish Thoracic Society (mBTS)，CURB65 et al. rules identifies patients with severe pneumonia but not patients who might be suitable for home management. A multicentre prospective study was conducted to derive and validate a practical severity assessment model for stratifying adults hospitalised with COVID-19 into different management groups.

DETAILED DESCRIPTION:
1. Screening interested participants should sign the appropriate informed consent (ICF) prior to completion any study procedures.
2. The investigator will review symptoms, risk factors, and other non-invasive inclusion and exclusion criteria.
3. The following is the general sequence of events during the 30-day evaluation period:
4. Completion of baseline procedures Participants were assessed for 30 days and completed all safety monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with novel coronavirus infection meeting the criteria of The New Coronavirus Pneumonia Diagnosis and Treatment Program (Ninth Edition);
2. Participants are willing to participate in this study and follow the research plan;
3. Participants or legally authorized representatives can give written informed consent approved by the Ethics Review Committee that manages the website.

Exclusion Criteria:

1. pneumonia was (a) not the primary cause for hospital admission, (b) an expected terminal event,or (c) distal to bronchial obstruction;
2. patients with tuberculosis,bronchiectasis,solid organ and haematological malignancies or human immuno deﬁciency virus (HIV) infection;
3. patients who had been in hospital within the previous 14days, were immunocompromised,or had previously been entered in the study;
4. nursing home residents.Participation in other clinical study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with novel coronavirus infection meeting the criteria of The New Coronavirus Pneumonia Diagnosis and Treatment Program (Ninth Edition)
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30days
  Mortality within 30days after diagnosis; Death from any cause
Deterioration of the condition | Day 1 to 30 days
  Deterioration of the condition: refer to Guidelines for the Diagnosis and Treatment of Novel Coronavirus Infection by the National Health Commission (Trial Version 9) The development from asymptomatic to mild/general-type. The development from mild to general-type/severe type The development from general-type to severe/critical type The development from severe to critical type

SECONDARY OUTCOMES:
Time to sustained disappearance of clinical symptoms | Up to 30 days
  Time to sustained disappearance of clinical symptoms
Percentage of participants with no clinical symptom | Day 3, 5, 7, 10, 14, 21 and 28
  Percentage of participants with no clinical symptoms from baseline to Day 3, 5, 7, 10, 14, 21 and 28
Percentage of participants who turned negative for SARS-CoV-2 and/or COVID-19 antigen | Day 3, 5, 7, 10, 14, 28
  Percentage of participants who turned negative for SARS-COV-2 COVID-19 antigen at Day 3, 5, 7, 10, 14, 28
Safety assessment Results: such as AEs and SAEs through Day 30 | Up to 30 days
  Safety assessment Results: such as AEs and SAEs through Day 30

CONTACTS AND LOCATIONS:
Overall Officials: zongyang yu, Ph.D, Principal Investigator — The 900th Hospital of the Joint Logistic Support Force, PLA
Locations (1):
- The 900th Hospital of the Joint Logistic Support Force, PLA, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ledford H. How severe are Omicron infections? Nature. 2021 Dec;600(7890):577-578. doi: 10.1038/d41586-021-03794-8. No abstract available. PMID 34934198
- [Result] Burki TK. Omicron variant and booster COVID-19 vaccines. Lancet Respir Med. 2022 Feb;10(2):e17. doi: 10.1016/S2213-2600(21)00559-2. Epub 2021 Dec 17. No abstract available. PMID 34929158
- [Result] Kupferschmidt K. Where did 'weird' Omicron come from? Science. 2021 Dec 3;374(6572):1179. doi: 10.1126/science.acx9738. Epub 2021 Dec 2. No abstract available. PMID 34855502
- [Result] Li Q, Nie J, Wu J, Zhang L, Ding R, Wang H, Zhang Y, Li T, Liu S, Zhang M, Zhao C, Liu H, Nie L, Qin H, Wang M, Lu Q, Li X, Liu J, Liang H, Shi Y, Shen Y, Xie L, Zhang L, Qu X, Xu W, Huang W, Wang Y. SARS-CoV-2 501Y.V2 variants lack higher infectivity but do have immune escape. Cell. 2021 Apr 29;184(9):2362-2371.e9. doi: 10.1016/j.cell.2021.02.042. Epub 2021 Feb 23. PMID 33735608
- [Result] Garcia-Beltran WF, Lam EC, St Denis K, Nitido AD, Garcia ZH, Hauser BM, Feldman J, Pavlovic MN, Gregory DJ, Poznansky MC, Sigal A, Schmidt AG, Iafrate AJ, Naranbhai V, Balazs AB. Multiple SARS-CoV-2 variants escape neutralization by vaccine-induced humoral immunity. Cell. 2021 Apr 29;184(9):2372-2383.e9. doi: 10.1016/j.cell.2021.03.013. Epub 2021 Mar 12. PMID 33743213
- [Result] Cao Y, Yisimayi A, Bai Y, Huang W, Li X, Zhang Z, Yuan T, An R, Wang J, Xiao T, Du S, Ma W, Song L, Li Y, Li X, Song W, Wu J, Liu S, Li X, Zhang Y, Su B, Guo X, Wei Y, Gao C, Zhang N, Zhang Y, Dou Y, Xu X, Shi R, Lu B, Jin R, Ma Y, Qin C, Wang Y, Feng Y, Xiao J, Xie XS. Humoral immune response to circulating SARS-CoV-2 variants elicited by inactivated and RBD-subunit vaccines. Cell Res. 2021 Jul;31(7):732-741. doi: 10.1038/s41422-021-00514-9. Epub 2021 May 21. PMID 34021265
- [Result] Pulliam JRC, van Schalkwyk C, Govender N, von Gottberg A, Cohen C, Groome MJ, Dushoff J, Mlisana K, Moultrie H. Increased risk of SARS-CoV-2 reinfection associated with emergence of Omicron in South Africa. Science. 2022 May 6;376(6593):eabn4947. doi: 10.1126/science.abn4947. Epub 2022 May 6. PMID 35289632
- [Result] Zhang X, Wu S, Wu B, Yang Q, Chen A, Li Y, Zhang Y, Pan T, Zhang H, He X. SARS-CoV-2 Omicron strain exhibits potent capabilities for immune evasion and viral entrance. Signal Transduct Target Ther. 2021 Dec 17;6(1):430. doi: 10.1038/s41392-021-00852-5. No abstract available. PMID 34921135